CLINICAL TRIAL: NCT02777866
Title: LAW Trial -The Impact of Local Anesthetics Infiltration in Surgical Wound of Gastrointestinal Procedures: A Blind Prospective Randomized Trial
Brief Title: LAW Trial -The Impact of Local Anesthetics Infiltration in Surgical Wound of Gastrointestinal Procedures
Acronym: LAW
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Noel Salgado Nesme, MD, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CIBH-1566
Record Dates: First submitted 2016-05-16; First posted 2016-05-19 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-04

CONDITIONS: Surgical Site Infection; Wound Infection; Postoperative Pain; Local Anesthetics
MeSH Terms: conditions — Surgical Wound Infection; Wound Infection; Pain, Postoperative | interventions — Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1: Bupivacaine 0.5% (Experimental): Patients who will be non urgent operated of an open gastrointestinal surgery, where an opening of the gastrointestinal lumen occurs (bile duct, stomach, small bowel or colon), who will be infiltrated in the total thickness of the abdominal wall (Peritoneum-muscle fascia- Subcutaneous tissue) with 0.5% Bupivacaine, every 1 cm, on each side of the surgical wound
  Interventions: Drug: Infiltration of 0.5% Bupivacaine
- 2: 0.9% Saline Solution (Placebo Comparator): Patients who will be non urgent operated of an open gastrointestinal surgery, where an opening of the gastrointestinal lumen occurs, who will be infiltrated in the total thickness of the abdominal wall with 0.9% Saline Solution, every 1 cm, on each side of the surgical wound.
  Interventions: Drug: Placebo: Infiltration of 0.9% Saline Solution

INTERVENTIONS:
Drug: Infiltration of 0.5% Bupivacaine — Patients who will be non urgent operated of an open gastrointestinal surgery, where an opening of the gastrointestinal lumen occurs (bile duct, stomach, small bowel or colon), who will be infiltrated in the total thickness of the abdominal wall (Peritoneum-muscle fascia- Subcutaneous tissue) with 0.5% Bupivacaine, every 1 cm, on each side of the surgical wound
  Arms: 1: Bupivacaine 0.5%
Drug: Placebo: Infiltration of 0.9% Saline Solution — Patients who will be non urgent operated of an open gastrointestinal surgery, where an opening of the gastrointestinal lumen occurs (bile duct, stomach, small bowel or colon), who will be infiltrated in the total thickness of the abdominal wall (Peritoneum-muscle fascia- Subcutaneous tissue) with 0.9% Saline Solution, every 1 cm, on each side of the surgical wound
  Arms: 2: 0.9% Saline Solution

SUMMARY:
The purpose of this study is to determine if the infiltration of 0.5% Bupivacaine in the surgical wound is effective to diminish the pain and the risk of surgical site infections in patients who go to a open gastrointestinal procedure.

DETAILED DESCRIPTION:
This is an experimental, randomized, prospective, double blind study, in which will compare two groups. First group of participants who will be non urgent operated of an open gastrointestinal surgery, where an opening of the gastrointestinal lumen occurs (bile duct, stomach, small bowel or colon), who will be infiltrated in the total thickness of the abdominal wall (Peritoneum-muscle fascia- Subcutaneous tissue) with 0.5% Bupivacaine, every 1 cm, on each side of the surgical wound; Second group of participants who will be non urgent operated of an open gastrointestinal surgery, where an opening of the gastrointestinal lumen occurs, who will be infiltrated in the total thickness of the abdominal wall with 0.9% Saline Solution, every 1 cm, on each side of the surgical wound.

In all participants undergoing to the protocol will make basic maneuvers to decreasing surgical site infection, which has already been standardized in the Institute. These maneuvers consist of administering prophylactic antibiotic 30 minutes before the incision, shaving of the abdominal wall with clipper in the OR, preoperative skin preparation with chlorhexidine gluconate 4%. All participants will get glucose control (<200 mg / dL), maintenance of the normothermia by putting hot air in the areas not exposed to the surgery field, heating fluids and getting intraoperative hyperoxia. Blood and components will be avoided as possible.

At the moment of closing of the abdominal wall, all the surgical personal will change the surgical gloves, also all the material that will be used should be sterile. The surgical nurse will pass the solution that will be injected, the investigator will not know the contents. 1 ml of the solution will be applied for each centimeter of the wound, covering the total thickness of the wall, on each side of the wound. After the closure of the fascia, the subcutaneous tissue will be washed with 1 liter of 0.9% saline solution. The skin will be closed with metal skin staples. The total administered dose of Bupivacaine should not be greater than stated as toxic (3mg/kg).

In all participants a 0.9% saline with 200 mg of Tramadol will be indicated for 24 hours. Participants may also receive IV Tramadol bolus of 25 mg, with a maximum of 4 in a day (top dose of 300 mg/day); in those participants in whom analgesia fails to control, the investigator may use other drugs like morphine of NSAIDs. No epidural or subarachnoid analgesia will be used.

All participants will be assessed 2 times per day for the presence of pain, this will be done with a numerical verbal scale from 0 to 10, when 0 is none pain, and 10 is the greatest pain that can reaches. The investigator will review the surgical wound once daily. The participant will be assessed every 7 days once discharged from hospital, in the outpatient clinic, until 30 days after the surgical procedure.

The sample size was calculated based on the incidence of surgical site infections in the Institute, which is 5%. The sample side required to demonstrate an expected reduction of 5% to 1%, with a power of 80% and a type 1 error of 5%, is 285 participants per group.

Randomization will be done electronically, which will be assigned 285 participants in each group.The investigators will annotate the number that will be given by the program in the participant expedient. The list of the numbers will be blind for investigators, and only the attending anesthesiologists will have it. The attending or resident anesthesiologist will give the syringe with the contents, being a blind study for the investigator and participant.

Statistical analysis will be performed using SPSS version 20.0 IBM, Microsoft Excel and numbers of iWorks for Macintosh. Statistical analysis according to the type of scaling of the variables analyzed will be performed. For comparison of dimensional variables will make a Student t test and ANOVA. For categorical variables a test of Kendall tau and chi square will be performed. Investigators will consider statistically significant any value equal or less than 0.05 or 5% for a hypothesis test two-tailed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are planned to a elective gastrointestinal surgery.
* Biliary-pancreatic open procedures: biliodigestive Derivation, Pancreatoduodenectomy, Pancreato-jejunostomy (Puestow procedure, Frey).
* Open upper gastrointestinal procedures: total gastrectomy, subtotal gastrectomy (distal gastrectomy with Billroth I reconstruction or Billroth II or Roux-Y), Gastro-jejunum anastomosis, Open gastro-jejunal Roux Y bypass, intestinal resection, intestinal reconnection, intestinal Fistulectomy.
* Open colorectal procedures: Right or Left Hemicolectomy, total colectomy, low anterior resection, abdominal-perineal resection.
* Patients who decide signing the informed consent after explained the study.
* Patients with postoperative follow-up of at least 30 days, in whom the wound and / or local complications will be evaluated.

Exclusion Criteria:

* Patients operated laparoscopically.
* Patients operated at another hospital.
* Patients with clean surgical wounds.
* Patients in whom an epidural or subarachnoid block is used.
* Patients who are unable to sign the informed consent.
* Patients with less than 50 kg.
* Patients wiht history of: Malignant hyperthermia, cardiac disease (Heart failure, history of myocardial infarction, arrhythmias), Epilepsy, Allergic to amides.
* Patients with incomplete follow-up (less than 30 days).
* Pregnant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 570 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Surgical Site Infection (SSI) defined by the Centre for Disease Control (CDC) criteria | 30 days following operation
  Postoperative surgical site infection (SSI), as defined by the following Centre for Disease Control (CDC) criteria:
  Infection occurring within the first 30 post-operative days with at least one of the following:
  1. Purulent drainage from the incision
  2. Organisms isolated from an aseptically obtained culture of fluid or tissue from the incision
  3. At least one of the following signs/symptoms of infection
     * Pain or tenderness
     * Localized swelling
     * Redness
     * Heat AND incision is deliberately opened by a surgeon (unless incision is culture negative)
  4. Diagnosis of SSI by the surgeon or attending physician
Efficacy of 0.5% Bupivacaine Infiltration for Post-op Pain measured using a Numeric Scale; 0-10 | Baseline to 48 hours postoperative
  Measurement of the efficacy of 0.5% Bupivacaine wound infiltration for the treatment of postoperative pain as measured by patient pain intensity (Numeric Scale; 0-10).

CONTACTS AND LOCATIONS:
Overall Officials: Noel Salgado-Nesme, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Tlalpan, Mexico City, Mexico City, Mexico